CLINICAL TRIAL: NCT01930344
Title: Does Three-Dimensional Laparoscopy Provide Significant Advantages for Patients and Surgeons? A Randomised Controlled Trial Investigating Operating Time and Surgical Errors With 3D vs 2D Visual Systems in Laparoscopic Cholecystectomies.
Brief Title: Investigating Three-Dimensional Versus Two-Dimensional Imaging in Laparoscopic Cholecystectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Katie Schwab MBBS BSc MRCS, Surgical Registrar & Research Fellow to MATTU, Royal Surrey County Hospital NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 13SURN0004; 13/EM/0092 (Other: UK Ethics Committee Reference)
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Gall Bladder Disease
Keywords: stereopsis; 3D laparoscopy; OCHRA
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3D laparoscopic visual system (Active Comparator): Laparoscopic cholecystectomy to be performed with 3D laparoscopic imaging system
  Interventions: Device: 3D Laparoscopic visual system
- 2D Laparoscopic Visual System (Placebo Comparator): Laparoscopic cholecystectomy to be performed using normal, 2D, laparoscopic visual system
  Interventions: Device: 2D Laparoscopic visual system

INTERVENTIONS:
Device: 3D Laparoscopic visual system — Three-dimensional endoscope used for surgery - multiple company products - and passive polarising three-dimensional laparoscopic displays;
  Arms: 3D laparoscopic visual system
Device: 2D Laparoscopic visual system — Standard 2D HD Laparoscopic Visual System
  Arms: 2D Laparoscopic Visual System

SUMMARY:
During laparoscopic surgery, your surgeon operates through 'keyhole' incisions in your abdomen. These allow long tools and a camera to pass to perform the surgery and allow the surgeon to see inside you. The cameras images are seen on a television screen, and this is viewed, like you watch television at home, in a two-dimensional (2D), form. This can make performing laparoscopic surgery very challenging, as you have to learn to appreciate depth while performing surgical tasks. Recent advances in viewing technology mean we now have the capability for comfortable three-dimensional (3D) viewing of laparoscopic surgery, and many centers have shown its superiority over 2D in lab-based experiments. However, this technology has never been compared against our normal gold standard 2D imaging in laparoscopic operations. This study aims to investigate whether there is a quantifiable benefit in using these new 3D imaging systems over 2D for laparoscopy, as we hypothesise that there is a marked benefit using 3D over 2D. Patients who have been placed on the waiting list for keyhole surgery to remove their gallbladder will be invited to take part in the study. If they agree, they will undergo the standard operation for removing their gallbladder as planned already. At the beginning of the operation they will be randomised (selected by chance) into one of two groups. One group will have their surgery performed to our current 'Gold standard' with the surgeon using a 2D camera and screen. The other group will have the exact same operation but with the surgeon using a 3D camera and screen. The intra-abdominal part of the operation will be recorded and viewed by an independent observer who is a surgeon, to assess for technical performance differences between operations performed in 2D and 3D, as well as time taken for the surgery. There are no extra risks to taking part and being randomised to the 3D group. The laparoscopic camera is the same size as a 2D camera and used in the same way. There are no real disadvantages, as patients will still undergo the operation they were booked for and will experience no change in their treatment. The aim is to compare 2D and 3D Day Case Laparoscopic Cholecystectomies, to see if there is a marked difference with this new technology. Lab based studies imply that 3D imaging systems reduce surgical errors and operating time therefore could improve patient safety. This study may help improve laparoscopic surgery for future patients.

DETAILED DESCRIPTION:
Laparoscopic surgery has been shown to improve patient recovery from surgical intervention, however it has a significant learning curve. This is related to the technical obstacles that need to be overcome and visually, losing the depth perception that accompanies its two- dimensional imaging. The advent of Robotic Surgery has demonstrated technical advantages due to the wristed instruments and three-dimensional imaging ability. The 3D vision or stereopsis of the robot significantly improves surgical performance, independently of the robotic tool advantages. Early investigators of three-dimensional imaging systems versus classical laparoscopic surgery did not demonstrate any significant benefit. This is likely to be related to the imaging capture and projection technology, which caused significant discomfort and eyestrain to the operator. In the last few years, there have been enormous leaps into the world of 3D vision and technology, associated with the film industry. Now 3D can be appreciated by mass audiences using polarising glasses that are simple to wear, without causing intolerable side-effects. The use of 3D technology has been compared with classical laparoscopy in many lab-based experiments and has shown to reduced technical errors and time of skill acquisition in trainees. These lab-based tests have also been completed by expert surgeons as part of PhD project undertaken by our previous research fellow, and although the data is unpublished yet, the results showed a 35% reduction in time and 60% reduction in errors in tests performed in 3D vs 2D. It is possible that 3D imaging will reduce operating time and improve patient safety in the operating theatre. We will be applying this research to true operations to show whether there is transference of these beneficial outcomes. With regard to surgical error, the assessment of surgical performance has led to several techniques which have been validated in the literature. We intend to utilise Human Reliability Analysis tools for the assessment of surgical error. The aim of this study is to address whether such a significant difference in performance will be observed in true surgery with these advances in 3D technology. This will be done by objectively assessing technical errors and operative time during routine gallbladder operations performed in 2D and 3D. There is no pilot study data, we are using the lab-based studies for the basis of calculations of power for numbers to be enrolled in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Listed for elective day case laparoscopic cholecystectomy

Exclusion Criteria:

* Previous upper abdominal surgery
* Significant previous gallbladder or pancreatic disease
* Unable to consent (due to cultural, language or neurological barriers)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Time of surgery | Measured at time of surgery
  Primary outcome is time of completion of the defined three steps of the operation, which is measured from the recorded video of the surgery.

SECONDARY OUTCOMES:
Errors enacted | Assessed from video recording of the surgery
  Two consultant surgeons, blinded to whether the surgery has been performed with 3D or 2D visual systems, will review the videos of the operations - edited to show 3 defined steps of surgery - to analyse for errors enacted by the operating surgeon. (Using the Observational clinical human reliability analysis, OCHRA, scoring system for error analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Rockall, MBBS MD, Study Chair — MATTU at Royal Surrey County Hospital, Guildford; Iain Jourdan, MA Mchir, Study Director — MATTU at Royal Surrey County Hospital, Guildford; Katie E Schwab, MBBS BSc, Principal Investigator — MATTU at Royal Surrey County Hospital, Guildford
Locations (1):
- Royal Surrey County Hospital, Guildford, Surrey, United Kingdom

REFERENCES:
- [Background] Hanna GB, Shimi SM, Cuschieri A. Randomised study of influence of two-dimensional versus three-dimensional imaging on performance of laparoscopic cholecystectomy. Lancet. 1998 Jan 24;351(9098):248-51. doi: 10.1016/S0140-6736(97)08005-7. PMID 9457094
- [Background] Jourdan IC, Dutson E, Garcia A, Vleugels T, Leroy J, Mutter D, Marescaux J. Stereoscopic vision provides a significant advantage for precision robotic laparoscopy. Br J Surg. 2004 Jul;91(7):879-85. doi: 10.1002/bjs.4549. PMID 15227695
- [Background] Smith R, Day A, Rockall T, Ballard K, Bailey M, Jourdan I. Advanced stereoscopic projection technology significantly improves novice performance of minimally invasive surgical skills. Surg Endosc. 2012 Jun;26(6):1522-7. doi: 10.1007/s00464-011-2080-8. Epub 2012 Jan 11. PMID 22234585
- [Background] McLachlan G. From 2D to 3D: the future of surgery? Lancet. 2011 Oct 15;378(9800):1368. doi: 10.1016/s0140-6736(11)61597-3. No abstract available. PMID 22010263
- [Background] Storz P, Buess GF, Kunert W, Kirschniak A. 3D HD versus 2D HD: surgical task efficiency in standardised phantom tasks. Surg Endosc. 2012 May;26(5):1454-60. doi: 10.1007/s00464-011-2055-9. Epub 2011 Dec 17. PMID 22179446
- [Background] Gurusamy KS, Sahay S, Davidson BR. Three dimensional versus two dimensional imaging for laparoscopic cholecystectomy. Cochrane Database Syst Rev. 2011 Jan 19;(1):CD006882. doi: 10.1002/14651858.CD006882.pub2. PMID 21249683
- [Background] Joice P, Hanna GB, Cuschieri A. Errors enacted during endoscopic surgery--a human reliability analysis. Appl Ergon. 1998 Dec;29(6):409-14. doi: 10.1016/s0003-6870(98)00016-7. PMID 9796785
- [Background] Miskovic D, Ni M, Wyles SM, Parvaiz A, Hanna GB. Observational clinical human reliability analysis (OCHRA) for competency assessment in laparoscopic colorectal surgery at the specialist level. Surg Endosc. 2012 Mar;26(3):796-803. doi: 10.1007/s00464-011-1955-z. Epub 2011 Nov 1. PMID 22042584
- [Background] Tang B, Hanna GB, Joice P, Cuschieri A. Identification and categorization of technical errors by Observational Clinical Human Reliability Assessment (OCHRA) during laparoscopic cholecystectomy. Arch Surg. 2004 Nov;139(11):1215-20. doi: 10.1001/archsurg.139.11.1215. PMID 15545569
- [Background] LaGrange CA, Clark CJ, Gerber EW, Strup SE. Evaluation of three laparoscopic modalities: robotics versus three-dimensional vision laparoscopy versus standard laparoscopy. J Endourol. 2008 Mar;22(3):511-6. doi: 10.1089/end.2007.0241. PMID 18269320
- [Derived] Schwab KE, Curtis NJ, Whyte MB, Smith RV, Rockall TA, Ballard K, Jourdan IC. 3D laparoscopy does not reduce operative duration or errors in day-case laparoscopic cholecystectomy: a randomised controlled trial. Surg Endosc. 2020 Apr;34(4):1745-1753. doi: 10.1007/s00464-019-06961-1. Epub 2019 Jul 16. PMID 31312963